CLINICAL TRIAL: NCT06468618
Title: Developing Restful Environments and Management Strategies for Pediatric Stem Cell Transplant Patients
Acronym: DREAMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Eric Zhou, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-254
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Stem Cell Transplant Complications; Sleep Disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DREAMS Program (Experimental): Enrolled participants and parent(s) will complete:
  * Baseline visit with survey
  * Standard of care stem cell infusion
  * In-clinic visit with introduction to DREAMS program, Sleep and Circadian Care Kit, Actigraph, and Fitbit.
  * Follow up survey
  Interventions: Behavioral: DREAMS Program Video and Care Kit

INTERVENTIONS:
Behavioral: DREAMS Program Video and Care Kit — A pediatric, circadian health program comprised of an introductory video to sleep experiences for stem cell transplant recipients, strategies to improve sleep, and a Sleep and Circadian Care Kit which includes ear plugs, a white noise machine, an eye mask, a lightbox, and kit instructions. Actigraph, Fitbit, and tablet will be provided to participant and family.

SUMMARY:
Pediatric patients undergoing stem cell transplant (SCT) are hospitalized for extended periods and are at high risk for sleep disturbances. In order to begin to address the environmental issues that SCT recipients face during inpatient hospitalizations, investigators will conduct a single arm pilot study of a program entitled 'Developing Restful Environments and Management Strategies' (DREAMS). The program will provide children receiving SCT and families with information and a kit that includes tools which may support sleep and circadian health during an inpatient hospitalization.

DETAILED DESCRIPTION:
In prior work, investigators conducted a study in which sound and light levels were recorded at one-minute intervals within an inpatient room on the SCT unit at Boston Children's Hospital using noise and light meters. Results showed that pediatric SCT recipients were consistently exposed to disruptive noise and light. Nighttime noise levels always exceeded World Health Organization recommendations for sleep, with recipients regularly exposed to multiple noise spikes associated with night wakings. While light levels were frequently dim enough to be conducive to sleep at night, participants were rarely exposed to light bright enough to preserve a healthy circadian rhythm during the day, which has the potential to dysregulate sleep at night. As a child's circadian rhythms may be affected by evening light to a greater extent than adults, such light spikes may be particularly disruptive to circadian rhythms in pediatric participants. The relatively low and afternoon-skewed daytime light, combined with the brighter than recommended light during the evening and early night, has been associated with longer hospitalizations and higher morbidity among adults.

This is a single-arm pilot study to evaluate the acceptability and feasibility of the DREAMS intervention program in stem cell transplant pediatric participants to help support families during this critical phase in a participant's SCT recovery. The data collected from this study will help understand the practicality of delivering the program to a greater number of participants and conducting clinical research about the program in the setting in which it will be implemented.

The research study procedures include screening for eligibility and surveys.

Participation in this research study is expected to last for about 2 weeks.

It is expected that about 10 children will take part in this research study.

The American Cancer Society is supporting this research study with grant funding.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 9-17 years.
* Patient scheduled to receive a stem cell transplant at Boston Children's Hospital.
* English speaking child and primary caregiver (parent/guardian).

Exclusion Criteria:

-Primary team declines permission to approach.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Enrollment Rate | Screening (Day -30 to -1)
  Defined as the proportion of eligible participants approached by research staff and consent to participate in the study with the cutoff set at ≥30% of eligible participants that are approached and agree to participate.
Acceptability of Intervention Measure Scale Score | At Follow-up Assessment Visit (Day 21, up to Day 28)
  Participants reporting an average score of ≥4 ("Agree") on the Acceptability of Intervention Measure scale, a four-item questionnaire assessing the acceptability of an intervention, on a 5-point scale with options ranging from Completely Agree to Completely Disagree.
DREAMS Care Kit Usage Rate | At Follow-up Assessment Visit (Day 21, up to Day 28)
  Feasibility of the DREAMS Program intervention is defined as ≥50% of participants reporting usage of at least one of the Care Kit materials.
Intervention Assessment Completion Rate | At Follow-up Assessment Visit (Day 21, up to Day 28)
  Feasibility of the DREAMS Program intervention is defined as ≥80% of enrolled participants completing the Follow-up Assessment.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Questionnaire | Baseline and Follow-up Assessment Visit (Day 21, up to Day 28)
  An 8-item measure used to assess the extent of a child's poor sleep. The minimum score is 8, and the maximum score is 40. Higher scores indicate worse sleep disturbance outcomes.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Questionnaire | Baseline and Follow-up Assessment Visit (Day 21, up to Day 28)
  An 8-item measure used to assess the extent of the consequences of a child's poor sleep. he minimum score is 8, and the maximum score is 40. Higher scores indicate worse sleep disturbance outcomes.
Sleep Diary | Daily, for 1 week, during the study period.
  A self-report of a participant's daily sleep patterns, including bedtime and total sleep duration.
Program Experience | At Follow-up Assessment Visit (Day 21, up to Day 28)
  Open-ended questions regarding what was liked/disliked about the Care Kit materials.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Zhou, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Background] Fidler AL, Waitt J, Lehmann LE, Solet JM, Duffy JF, Gonzalez BD, Beebe DW, Fedele DA, Zhou ES. Sleep and circadian disruptors: Unhealthy noise and light levels for hospitalized pediatric patients. J Hosp Med. 2023 Nov;18(11):999-1003. doi: 10.1002/jhm.13218. Epub 2023 Oct 2. PMID 37779507